CLINICAL TRIAL: NCT05353946
Title: CRATER Trial: Coronary Rotational Atherectomy Elective vs. Bailout in Patients With Severely Calcified Lesions and Chronic Renal Failure
Brief Title: Coronary Rotational Atherectomy Elective vs. Bailout in Severely Calcified Lesions and Chronic Renal Failure
Acronym: CRATER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guillermo Galeote; MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Guillermo Galeote; MD, PhD, Principal Investigator, Hospital Universitario La Paz
Organization: Hospital Universitario La Paz (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00001
Record Dates: First submitted 2022-04-06; First posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Coronary Artery Disease; Chronic Renal Failure
Keywords: Severely calcified coronary lesion; Rotational atherectomy; Chronic kidney disease; Intravascular ultrasound; Percutaneous coronary intervention
MeSH Terms: conditions — Coronary Artery Disease; Kidney Failure, Chronic; Renal Insufficiency, Chronic | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Elective Rotational Atherectomy (Active Comparator): Operators can decide elective use of rotational atherectomy (RA) or conventional angioplasty according to the calcification patterns of the coronary lesion evaluated by Intravascular ultrasound (IVUS) or by angiography if the IVUS cannot cross the lesion.
  Procedure is performed with a Rotablator system, consisting of a rotating olive-shaped burr whose leading hemisphere is coated with microscopic diamond chips. The proximal end of the device has a housing unit containing the burr advancer, a fiberoptic tachometer cable, an irrigation port, and a nitrogen gas delivery hose, which permits the rapidly rotating of the burr. The RA catheter is introduced into the coronary artery over a stainless steel 0.09-inch wire to cross the lesion, then advanced with a slow pecking motion at a speed of 160,000 to 190,000 rpm with each ablation run <15 seconds is performed. Burr size was with a burr/vessel ratio of 0.7. After RA, all patients received IVUS-guided percutaneous coronary intervention.
  Interventions: Device: Percutaneous coronary intervention (PCI)
- Bailout Rotational Atherectomy (Active Comparator): The operators began with conventional angioplasty (non-compliant balloon dilatation) regardless of the calcification patterns in the coronary lesion, and rotational atherectomy (RA) can be used only as a bailout.
  Interventions: Device: Percutaneous coronary intervention (PCI)

INTERVENTIONS:
Device: Percutaneous coronary intervention (PCI) — Optimal stent expansion by IVUS-guided PCI.

SUMMARY:
The current role of the rotational atherectomy is for non-dilatable coronary lesions and for severely calcified lesions that may interfere with optimal stent expansion.

Severely calcified coronary lesions are associated with worse outcomes. In this regard, chronic kidney disease is associated with severely calcified coronary arteries.

Some evidence suggests that elective rotational atherectomy used by experienced operators can be safe and effective, minimizing time and complications for patients with heavily calcified lesions.

However, there is no direct randomized comparison between rotational atherectomy and angioplasty alone in the setting of chronic renal failure and with intravascular ultrasound assessment for detecting severely calcified coronary arteries.

DETAILED DESCRIPTION:
The current role of the rotational atherectomy is for non-dilatable coronary lesions and for severely calcified lesions that may interfere with optimal stent expansion.

Severely calcified coronary lesions are associated with worse outcomes. In this regard, chronic kidney disease is associated with severely calcified coronary arteries.

Some evidence suggests that elective rotational atherectomy used by experienced operators can be safe and effective, minimizing time and complications for patients with heavily calcified lesions.

However, there is no direct randomized comparison between rotational atherectomy and angioplasty alone in the setting of chronic renal failure and with intravascular ultrasound assessment for detecting severely calcified coronary arteries.

The aim of this study is to compare the healthcare cost analysis between elective atherectomy and conventional atherectomy (bailout). The secondary endpoints were stent placement success (defined as expansion with <20% residual stenosis assessed by intravascular ultrasound and TIMI 3 flow without crossover or stent failure), procedure time, radiation exposure, periprocedural and in-hospital complications, and major cardiovascular adverse events at medium-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years.
* Glomerular filtration rate (GFR) <60 mL/min/1.73 m2 for 3 months or more
* Stenosis ≥70% in a coronary artery with a diameter ≥2,5 mm.
* Severe angiographic calcification (affecting both sides of the arterial lumen)
* Any clinical scenario except acute myocardial infarction in the first seven days of evolution.
* Native coronary vessel or bypass graft.

Exclusion Criteria:

* Absence of informed consent.
* Acute myocardial infarction in the first 7 days of evolution.
* Lesion in a single patent vessel.
* Calcified lesions with an angulation >60º, dissections, lesions with thrombus, and degenerated saphenous vein grafts.
* Hemodynamically unstable patients
* Patients with allergy to iodinated contrast media
* Patients with significant comorbidity and with a life expectancy of less than one year

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2019-02-02 (Actual); Primary Completion 2022-12-27 (Estimated); Study Completion 2023-12-04 (Estimated)

PRIMARY OUTCOMES:
The healthcare cost analysis between elective atherectomy and conventional atherectomy (bailout) | Periprocedural and 30 days after the procedure
  The costs included the items, supplies, and time used in the catheterization laboratory, and expenses caused by complications during hospital length of stay and 30 days after the procedure.

SECONDARY OUTCOMES:
The healthcare cost analysis between elective atherectomy and conventional atherectomy (bailout) | Follow-up 5 years.
  During follow-up 5 years.
Contrast-induced nephropathy | 48 hours after the procedure.
  Contrast-induced nephropathy 48 hours after the procedure.
Stent placement success | Periprocedural
  Defined as expansion with <20% residual stenosis assessed by intravascular ultrasound and TIMI 3 flow without crossover or stent failure
The amount of angioplasty balloons used in each group before stent deployment. | Periprocedural
  Number of semi-compliant and non-compliant balloons used during procedure deployment.
Procedure and fluoroscopy times | Periprocedural
  Measured in minutes
Periprocedural complications | Periprocedural
  Coronary dissection (NHLBI classification system), coronary perforation (Ellis classification system), no-reflow phenomenon (defined as less than TIMI 3 flow), and side branch occlusion
In-hospital complications | during hospitalization stay until discharge
  Target lesion revascularization, target vessel revascularization, non-target vessel revascularization, stent thrombosis, vascular complications, and death
Major cardiovascular events | 1,2,3,4 and 5 years after procedure
  Death, myocardial infarction, target lesion revascularization, target vessel revascularization, and non-target vessel revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Galeote, PhD, MD, Principal Investigator — La Paz University Hospital
Locations (1):
- La Paz University Hospital, Madrid, Spain